CLINICAL TRIAL: NCT04173494
Title: A Randomized, Double-blind, Phase 3 Study to Evaluate the Activity of Momelotinib (MMB) Versus Danazol (DAN) in Symptomatic, Anemic Subjects With Primary Myelofibrosis (PMF), Post-polycythemia Vera (PV) Myelofibrosis, or Post-essential Thrombocythemia (ET) Myelofibrosis Who Were Previously Treated With JAK Inhibitor Therapy
Brief Title: A Study of Momelotinib Versus Danazol in Symptomatic and Anemic Myelofibrosis Participants (MOMENTUM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRA-MMB-301
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: Myelofibrosis; JAK inhibitor; Danazol; Momelotinib; Functional Iron deficiency; Activin receptor type 1; Anemia; Transfusion; Hepcidin; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases
MeSH Terms: conditions — Primary Myelofibrosis; Anemia; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide; Danazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the 24 week randomized treatment phase of the study, participants, investigators and sponsor and relevant vendor personnel (with the exception of specified unblinded personnel, for example clinical supply) will remain blinded to the participant's treatment assignment and to aggregate data that may lead to inadvertent unblinding. Participants who continue treatment with momelotinib or danazol after Week 24 in the extended treatment phase will receive unblinded treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Momelotinib (Experimental): Participants will receive momelotinib plus placebo to match danazol
  Interventions: Drug: Momelotinib; Drug: Placebo to match danazol
- Danazol (Active Comparator): Participants will receive danazol plus placebo to match momelotinib
  Interventions: Drug: Danazol; Drug: Placebo to match momelotinib

INTERVENTIONS:
Drug: Momelotinib — Momelotinib tablets will be self-administered orally once daily
  Other Names: MMB, GS-0387, CYT387
  Arms: Momelotinib
Drug: Placebo to match danazol — Danazol placebo capsules will be self-administered orally twice daily
  Arms: Momelotinib
Drug: Danazol — Danazol capsules will be self-administered orally twice daily
  Other Names: Danocrine
  Arms: Danazol
Drug: Placebo to match momelotinib — Momelotinib placebo tablets will be self-administered orally once daily
  Arms: Danazol

SUMMARY:
MOMENTUM is a randomized, double-blind, active control Phase 3 trial intended to confirm the differentiated clinical benefits of the investigational drug momelotinib (MMB) versus danazol (DAN) in symptomatic and anemic participants who have previously received an approved Janus kinase inhibitor (JAKi) therapy for myelofibrosis (MF). The purpose of this clinical study is to compare the effectiveness and safety of MMB to DAN in treating and reducing: 1) disease related symptoms, 2) the need for blood transfusions and 3) splenomegaly, in adults with primary MF, post-polycythemia vera MF or post-essential thrombocythemia MF. The study is planned in countries including, but not limited to: Australia, Austria, Belgium, Bulgaria, Canada, Czech Republic, Denmark, France, Germany, Hungary, Israel, Italy, New Zealand, Poland, Romania, Singapore, South Korea, Spain, Sweden, Taiwan, United Kingdom (UK) and United States (US).

Participants must be symptomatic with a Myelofibrosis Symptom Assessment Form (MFSAF) version (v) 4.0 Total Symptom Score of >= 10 at screening, and be anemic with hemoglobin (Hgb) < 10 gram/deciliter (g/dL). For participants with ongoing JAKi therapy at screening, JAKi therapy must be tapered over a period of at least 1 week, followed by a 2-week non-treatment washout interval prior to randomization.

Participants will be randomized 2:1 to orally self-administer blinded treatment: MMB plus placebo or DAN plus placebo. Participants randomized to receive MMB who complete the randomized treatment period to the end of Week 24 may continue to receive MMB in the open-label extended treatment period to the end of Week 204 (a total period of treatment of approximately 4 years) if the participants tolerates and continues to benefit from MMB.

Participants randomized to receive DAN may cross-over to MMB open-label treatment in the following circumstances: at the end of Week 24 if they complete the randomized treatment period; or at the end of Week 24 if they discontinue treatment with DAN but continue study assessments and do not receive prohibited medications including alternative active anti-MF therapy; or at any time during the randomized treatment period if they meet the protocol-defined criteria for radiographically confirmed symptomatic splenic progression. Participants randomized to receive DAN who are receiving clinical benefit at the end of Week 24 may choose to continue DAN therapy up to Week 48. The comparator treatment, DAN, is an approved medication in the US and in some other countries and is recommended by national guidelines as a treatment for anemia in MF.

DETAILED DESCRIPTION:
MOMENTUM Contact Email: GSKClinicalSupportHD@gsk.com

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Confirmed diagnosis of PMF in accordance with the World Health Organization (WHO) 2016 criteria, or Post- polycythemia vera/essential thrombocythemia (PV/ET) MF in accordance with the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT criteria).
* Symptomatic, defined as a TSS of >= 10 units assessed by a single MFSAF v4.0 assessment during Screening prior to Baseline period (Day BL1).
* Anemic, defined as a Hgb < 10 g/dL in Screening/Baseline period.
* Previously treated with an approved JAK inhibitor for PMF or Post-PV/ET MF for >= 90 days, or >= 28 days if JAK inhibitor therapy is complicated by RBC transfusion requirement of >= 4 units in 8 weeks, or Grade 3/4 AEs of thrombocytopenia, anemia, or hematoma.
* Baseline splenomegaly, defined as having a palpable spleen at >= 5 centimeter (cm), below the left costal margin, or with volume >= 450 cubic centimeter (cm^3) on imaging (ultrasound, magnetic resonance imaging [MRI] or computed tomography [CT] are acceptable), assessed during Screening at any point prior to Randomization.
* High risk, intermediate-2, or intermediate-1 risk MF as defined by Dynamic International Prognostic Scoring System (DIPSS), or DIPSS-plus.
* No allogeneic stem cell transplant planned.
* Acceptable laboratory assessments:

  1. Absolute neutrophil count (ANC) >= 0.75 × 10^9/Liter (L).
  2. Platelet count (PLT) >= 25 × 10^9/L (without requirement for platelet transfusion).
  3. Peripheral blast count < 10%.
  4. Alanine aminotransferase/ glutamic-oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/ serum glutamic-pyruvic transaminase (ALT/SGPT) <= 3 × Upper Limit Normal (ULN) (<= 5 × ULN if liver is involved by extramedullary hematopoiesis as judged by the investigator or if related to iron chelator therapy that was started within the prior 60 days).
  5. Calculated creatinine clearance (CCr) >= 30 milliliter per minute (mL/min) according to Cockcroft-Gault.
  6. Direct bilirubin <= 2.0 × ULN.

Exclusion Criteria:

* Use of the following treatments within the time periods noted:

  1. Prior momelotinib treatment at any time.
  2. Approved JAK inhibitor therapy (eg, fedratinib or ruxolitinib) within 1 week prior to the first day of Baseline.
  3. Active anti-MF therapy within 1 week prior to the first day of Baseline.
  4. Potent Cytochrome P450 3A4 (CYP3A4) inducers within 1 week prior to Randomization.
  5. Investigational agent (including investigational JAK inhibitors) within 4 weeks prior to Randomization.
  6. Erythropoiesis stimulating agent (ESA) within 4 weeks prior to Randomization.
  7. Danazol within 3 months prior to Randomization.
  8. Splenic irradiation within 3 months prior to Randomization.
  9. Current treatment with simvastatin, atorvastatin, lovastatin or rosuvastatin.
* History of prostate cancer, with the exception of localized prostate cancer that has been treated surgically or by radiotherapy with curative intent and presumed cured.
* Prostate specific antigen (PSA) > 4 nanograms per milliliter (ng/mL).
* Unsuitable for spleen volume measurements due to prior splenectomy or unwilling or unable to undergo an MRI scan or CT scan for spleen volume measurement per protocol requirements.
* Any of the following (criteria a - k):

  1. Uncontrolled intercurrent illness including, but not limited to: active uncontrolled infection (participants receiving outpatient antibacterial and/or antiviral treatments for infection that is under control or as infection prophylaxis may be included in the trial).
  2. Significant active or chronic bleeding event >= Grade 2 per Common Terminology Criteria for Adverse Events (CTCAE) v5.0, within 4 weeks prior to Randomization.
  3. Unstable angina pectoris within 6 months prior to Randomization.
  4. Symptomatic congestive heart failure within 6 months prior to Randomization.
  5. Uncontrolled cardiac arrhythmia within 6 months prior to Randomization.
  6. QT Interval Corrected Using Fridericia's Formula (QTcF) interval > 500 millisecond (msec), unless attributed to bundle branch block.
  7. Current progressive thrombosis despite treatment.
  8. History of porphyria.
  9. Child-Pugh score >= 10.
  10. Psychiatric illness, social situation, or any other condition that would limit compliance with trial requirements or may interfere with the interpretation of study results, as judged by investigator or sponsor.
  11. Inability or unwillingness to comply with the protocol restrictions on MF therapy and other medications prior to and during study treatment.
* Participants with a prior or concurrent malignancy, whose natural history or treatment has a significant potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding or thalassemia.
* Known positive status for human immunodeficiency viruses (HIV).
* Chronic active or acute viral hepatitis A, B, or C infection, or hepatitis B or C carrier (testing required for hepatitis B and C).
* Unresolved non-hematologic toxicities from prior therapies that are > Grade 1 per CTCAE v5.0.
* Presence of peripheral neuropathy >= Grade 2 per CTCAE v5.0.
* Women who are already pregnant or lactating. Additional inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, M.D., Ph.D., Principal Investigator — Department of Leukemia, The University of Texas MD Anderson Cancer Center; Ruben Mesa, Principal Investigator — UT Health San Antonio Cancer Center, San Antonio, TX, USA
Locations (167):
- United States (17):
  - Mayo Clinic Hospital - Phoenix, Phoenix, Arizona
  - Irvine Center for Clinical Research, Irvine, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - American Institute of Research - Whittier, Whittier, California
  - University of Colorado Hospital Anschutz Cancer Pavilion, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Northwest Oncology & Hematology - Rolling Meadows, Rolling Meadows, Illinois
  - Washington University School of Medicine in Saint Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Irving Medical Center - Presbyterian Hospital, New York, New York
  - Cleveland Clinic - Richard E. Jacobs Health Center, Avon, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Australia (5):
  - Canberra Region Cancer Centre, Garran, Australian Capital Territory
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Perth Radiological Clinic - Magnetic Resonance Centre, Perth, Western Australia
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Ordensklinikum Linz Elisabethinen, Linz, Upper Austria
  - Medizinische Universität Wien, Vienna, Vienna
  - Oberösterreichische Gesundheitsholding GmbH, Steyr
- Belgium (5):
  - Hôpital Erasme, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi - Notre Dame, Charleroi, Hainaut
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Centre Hospitalier Universitaire de Liège, Liège
- Bulgaria (4):
  - University Multiprofile Hospital For Active Treatment Dr. Georgi Stranski EAD, Pleven
  - University Hospital St. Ivan Rilski, Sofia
  - University Multiprofile Hospital For Active Treatment Aleksandrovska, Sofia
  - National Specialized Hospital for Active Treatment of Haematologic Diseases, Sofia
- Canada (6):
  - Saint Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre - Halifax Infirmary, Halifax, Nova Scotia
  - McMaster University Medical Center, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Research Institute of the McGill University Health Centre, Montreal, Quebec
  - Hôpital de l'Enfant-Jésus, Québec
- Fakultni Nemocnice Brno, Brno, Jihormoravsky Kraj, Czechia
- Denmark (4):
  - Herlev Hospital, Herlev, Capital Region
  - Aalborg Universitetshospital - Syd, Aalborg, North Denmark
  - Sjællands Universitetshospital - Roskilde, Roskilde, Region Sjælland
  - Odense Universitetshospital, Odense, Region Syddanmark
- France (17):
  - Hôpital Haut-Lévêque, Pessac, Aquitaine
  - Hospital Center University Of Caen Normandie, Caen, Basse-Normandie
  - Hôpital Claude Huriez, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire Limoges, Limoges, Limousin
  - Centre Hospitalier De Lens, Lens, Nord Pas-Des-Calais
  - Centre Hospitalier Le Mans, Le Mans, Pays de la Loire Region
  - Centre Hospitalier Universitaire Amiens-Picardie - Site Sud, Amiens, Picardie
  - Hôpital l'Archet, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Rhone-Alps
  - Centre Hosptitalier Universitaire Angers, Angers
  - Hôpital Saint-Vincent De Paul - Lille, Lille
  - Hôpital De La Conception, Marseille
  - Hôpital Emile Muller, Mulhouse
  - Centre Hospitalier Universitaire Nantes - Hôtel Dieu, Nantes
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hôpital Saint-Louis, Paris, Île-de-France Region
  - Hôpital Saint-Antoine, Paris, Île-de-France Region
- Germany (10):
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Jena, Jena, Thuringia
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Kliniken Ostalb - Stauferklinikum Schwäbisch Gmünd, Mutlangen
- Hungary (9):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Szent Borbála Kórház, Tatabánya, Komárom-Esztergom
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet - Szent László Telephely, Budapest, Pest County
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Szabolcs-Szatmár-Bereg Megyei Kórházak És Egyetemi Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Markusovszky Egyetemi Oktatókórház Szombathely, Szombathely, Vas County
  - Semmelweis Egyetem, Budapest
  - Petz Aladár Megyei Oktató Kórház, Győr
- Israel (10):
  - Yitzhak Shamir Medical Center, Be’er Ya‘aqov, Central District
  - Bnai Zion Medical Center, Haifa, Haifa District
  - Hadassah University Hospital Ein Kerem, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Western Galilee Hospital-Nahariya, Nahariya
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (20):
  - Azienda Ospedaliero - Universitaria Careggi, Florence, Florence
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-Cesena
  - Azienda Socio Sanitaria Territoriale Monza - Ospedale San Gerardo, Monza, Monza E Brianza
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, Pesaro E Urbino
  - IRCCS Centro di Riferimento Oncologico di Basilicata, Rionero in Vulture, Potenza
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino, Turin
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino, Turin
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo - Alessandria, Alessandria
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna
  - Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Umberto I - Policlinico di Roma, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Presidio Ospedaliero Universitario Santa Maria della Misericordia, Udine
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale Policlinico Giambattista Rossi Borgo Roma, Verona
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Middlemore Clinical Trials, Auckland
- Poland (10):
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow, Lesser Poland Voivodeship
  - Klinika Hematologii Nowotworów Krwi i Transplantacji Szpiku, Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin, Lublin Voivodeship
  - Instytut Hematologii I Transfuzjologii, Warsaw, Masovian Voivodeship
  - Alvamed Zakład Specjalistycznej Opieki Zdrowotnej, Warsaw, Masovian Voivodeship
  - Szpital Wojewódzki w Opolu, Opole, Opole Voivodeship
  - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk, Pomeranian Voivodeship
  - Silesian Healthy Blood Clinic, Chorzów, Salskie
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Łodzi, Lodz
- Romania (5):
  - Spitalul Filantropia - Craiova, Craiova, Dolj
  - Institutul Regional De Oncologie Iasi, Iași, Iaşi
  - Spitalul Clinic Judetean De Urgenta Târgu Mureș, Târgu Mureş, Mureș County
  - Laboratul clinic MedLife-Policlinica de Diagnostic Rapid Brasov, Brasov
  - Coltea - Spital Clinic, Bucharest
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (9):
  - Kyungpook National University Hospital, Daegu, Daegu Gwang'yeogsi
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul Saint Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (13):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Institut Hospital del Mar d'Investigacions Mèdiques, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Institut Català d'Oncologia Girona, Girona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia
  - Hospital de Día Quirónsalud Zaragoza, Zaragoza
- Sweden (3):
  - Karolinska Universitetssjukhuset Solna, Solna, Stockholm County
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County
  - Uddevalla Sjukhus, Uddevalla
- Taiwan (4):
  - Chiayi Chang Gung Memorial Hospital, Buzi, Chaiyi
  - China Medical University Hospital, Taichung, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District
- United Kingdom (7):
  - United Lincolnshire Hospitals NHS Trust, Boston, England
  - University Hospitals Bristol NHS Foundation Trust, Bristol, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - Guy's and Saint Thomas' NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, England
  - NHS Lanarkshire, Airdrie, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon SS, Chen CC, Lee SE, Chang H, Cheong JW, Hou HA, Lee WS, Lim SN, Moon JH, Ong KH, Dai Y, Liu C, Kawashima J, Goh YT. Efficacy and safety of momelotinib in Janus kinase inhibitor-experienced Asian patients with myelofibrosis and anemia. Int J Hematol. 2025 Nov;122(5):660-670. doi: 10.1007/s12185-025-04037-6. Epub 2025 Jul 21. PMID 40691344
- [Derived] Mesa RA, Talpaz M, Mazerolle F, Gorsh B, M'Hari M, Regnault A, Ellis C, Wang Z, Purser M, Liu T, Strouse B, Patnaik D. Time Without Transfusion Reliance (TWiTR): Integrating Survival Quality Into Myelofibrosis Treatment Strategies Based on the Phase 3 SIMPLIFY-1, SIMPLIFY-2, and MOMENTUM Trials. EJHaem. 2025 Jun 18;6(3):e70075. doi: 10.1002/jha2.70075. eCollection 2025 Jun. PMID 40535755
- [Derived] Harrison CN, Mesa R, Talpaz M, Gupta V, Gerds AT, Perkins A, Goh YT, Fox ML, McLornan D, Palmer J, Foltz L, Vannucchi A, Koschmieder S, Passamonti F, Lee SE, Ellis C, Strouse B, Gonzalez Carreras FJ, Oh ST. Longitudinal Assessment of Transfusion Intensity in Patients With JAK Inhibitor-Naive or -Experienced Myelofibrosis Treated With Momelotinib. Clin Lymphoma Myeloma Leuk. 2025 Mar;25(3):199-211. doi: 10.1016/j.clml.2024.10.001. Epub 2024 Oct 16. PMID 39516087
- [Derived] Gerds AT, Verstovsek S, Vannucchi AM, Al-Ali HK, Lavie D, Kuykendall AT, Grosicki S, Iurlo A, Goh YT, Lazaroiu MC, Egyed M, Fox ML, McLornan D, Perkins A, Yoon SS, Gupta V, Kiladjian JJ, Granacher N, Lee SE, Ocroteala L, Passamonti F, Harrison CN, Oh S, Klencke BJ, Yu J, Donahue R, Kawashima J, Mesa R. Momelotinib versus danazol in symptomatic patients with anaemia and myelofibrosis previously treated with a JAK inhibitor (MOMENTUM): an updated analysis of an international, double-blind, randomised phase 3 study. Lancet Haematol. 2023 Sep;10(9):e735-e746. doi: 10.1016/S2352-3026(23)00174-6. Epub 2023 Jul 27. PMID 37517413
- [Derived] Verstovsek S, Mesa R, Gupta V, Lavie D, Dubruille V, Cambier N, Platzbecker U, Hus M, Xicoy B, Oh ST, Kiladjian JJ, Vannucchi AM, Gerds A, Egyed M, Mayer J, Sacha T, Kawashima J, Morris M, Huang M, Harrison C. Momelotinib long-term safety and survival in myelofibrosis: integrated analysis of phase 3 randomized controlled trials. Blood Adv. 2023 Jul 25;7(14):3582-3591. doi: 10.1182/bloodadvances.2022009311. PMID 37042865
- [Derived] Verstovsek S, Gerds AT, Vannucchi AM, Al-Ali HK, Lavie D, Kuykendall AT, Grosicki S, Iurlo A, Goh YT, Lazaroiu MC, Egyed M, Fox ML, McLornan D, Perkins A, Yoon SS, Gupta V, Kiladjian JJ, Granacher N, Lee SE, Ocroteala L, Passamonti F, Harrison CN, Klencke BJ, Ro S, Donahue R, Kawashima J, Mesa R; MOMENTUM Study Investigators. Momelotinib versus danazol in symptomatic patients with anaemia and myelofibrosis (MOMENTUM): results from an international, double-blind, randomised, controlled, phase 3 study. Lancet. 2023 Jan 28;401(10373):269-280. doi: 10.1016/S0140-6736(22)02036-0. PMID 36709073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the activity of Momelotinib (MMB) versus Danazol (DAN) in Symptomatic, Anemic participants. This study consists of Randomized Double-blind (DB) Treatment Period (TP) and Open-label extended Treatment Period.
Pre-assignment Details: A total of 195 participants were enrolled in the study.
Groups:
- MMB 200 mg Once Daily (QD) + Placebo: Participants were randomized to receive 200 milligrams (mg) of MMB orally QD and a DAN-placebo orally twice daily (BID) during the randomized 24-week double-blind treatment period. Participants who completed the randomized treatment period or discontinued treatment early for other reasons but completed scheduled assessments through Week 24 were enrolled in an open-label extended treatment period. Participants continued to receive 200 mg of MMB orally QD during the open-label extended treatment period. Participants who discontinued treatment prior to Week 24 due to splenic progression or other reasons, but completed assessments, were unblinded. Participants who discontinued MMB during the randomized treatment period were not eligible to receive MMB in the open-label extended treatment period. Participants who were randomized to MMB during the randomized treatment period with confirmed splenic progression could not proceed to the open-label extended treatment period.
- DAN 300 mg BID + Placebo: Participants were randomized to receive 300 mg of DAN orally BID and MMB-placebo orally QD during the randomized 24-week double-blind treatment period. Participants who completed the randomized treatment period, discontinued treatment early due to splenic progression, or discontinued treatment early for other reasons but completed scheduled assessments through Week 24 enrolled in an open-label extended treatment period. Participants switched to receive 200 mg of MMB orally QD during open-label extended treatment period. All participants elected to receive MMB as open-label treatment during the open-label extended treatment period.
Period: Randomized DB TP (Up to Week 24)
Arm/Group | MMB 200 mg Once Daily (QD) + Placebo | DAN 300 mg BID + Placebo
Started | 130 | 65
Completed | 94 | 38
Not Completed | 36 | 27
Not completed — Adverse Event | 16 | 11
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lack of Efficacy | 6 | 3
Not completed — Death | 4 | 3
Not completed — Leukemic Transformation | 2 | 2
Not completed — Disease Progression | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Open-Label Extended TP(Weeks 24 to 151)
Arm/Group | MMB 200 mg Once Daily (QD) + Placebo | DAN 300 mg BID + Placebo
Started | 93 (93 participants from Randomized Treatment Phase entered in Open-label Phase) | 41 (Total 41 participants entered in Open-label Phase (36 out of 38 participants who completed Randomized Phase and 5 out of 27 who withdrew from Randomized Phase) as per Protocol defined criteria.)
Completed | 0 | 0
Not Completed | 93 | 41
Not completed — Adverse Event | 11 | 1
Not completed — Death | 6 | 3
Not completed — Lack of Efficacy | 6 | 2
Not completed — Physician Decision | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Leukemic transformation | 0 | 1
Not completed — Disease progression | 1 | 1
Not completed — Continuing in MMB extension study | 61 | 27

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were measured in the Intention-To-Treat (ITT) Analysis Set, which included all randomized participants.
Groups:
- MMB 200 mg QD + Placebo: Participants were randomized to receive 200 milligrams (mg) of MMB orally QD and a DAN-placebo orally twice daily (BID) during the randomized 24-week double-blind treatment period. Participants who completed the randomized treatment period or discontinued treatment early for other reasons but completed scheduled assessments through Week 24 were enrolled in an open-label extended treatment period. Participants continued to receive 200 mg of MMB orally QD during the open-label extended treatment period. Participants who discontinued treatment prior to Week 24 due to splenic progression or other reasons, but completed assessments, were unblinded. Participants who discontinued MMB during the randomized treatment period were not eligible to receive MMB in the open-label extended treatment period. Participants who were randomized to MMB during the randomized treatment period with confirmed splenic progression could not proceed to the open-label extended treatment period.
- DAN 300 mg BID + Placebo: Participants were randomized to receive 300 mg of DAN orally BID and MMB-placebo orally QD during the randomized 24-week double-blind treatment period. Participants who completed the randomized treatment period, discontinued treatment early due to splenic progression, or discontinued treatment early for other reasons but completed scheduled assessments through Week 24 were enrolled in an open-label extended treatment period. Participants who received DAN 300 mg BID during randomized period switched to receive 200 mg of MMB orally QD during open-label extended treatment period.
- Total: Total of all reporting groups
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo | Total
Number analyzed (Participants) | 130 | 65 | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.85 (8.24) | 71.46 (6.99) | 70.38 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 21 | 72
  Male | 79 | 44 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 115 | 54 | 169
  Unknown or Not Reported | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 107 | 50 | 157
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Total Symptom Score (TSS) Response Rate at Week 24
Description: Myelofibrosis Symptom Assessment Form (MFSAF) TSS version (v) 4.0 response rate was defined as percentage of participants with a >= 50 percent (%) reduction from Baseline in mean MFSAF TSS over consecutive 28-day period immediately before end of Week 24. TSS response rate was measured using MFSAF v4.0. MFSAF v4.0 comprises 7 domains representing 7 most relevant symptoms of myelofibrosis (MF) identified through existing participant and clinician-based evidence: fatigue,night sweats,pruritus,abdominal discomfort,pain under left ribs,early satietyand bone pain. Participants scored each symptom domain using an 11-point numeric rating scale ranging from 0(absent) to 10(worst imaginable). The MFSAF TSS was calculated as sum of scores of 7 domains for a possible range of scores of 0 to 70, with a higher TSS corresponding to more severe symptoms. A reduction from Baseline corresponded to a lessening of MF symptoms. Baseline was the last assessment done before or on the day of first dose date.
Time Frame: Baseline and Week 24
Population: Measured in the Intent-To-Treat (ITT) Analysis Set, which included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Percentage of participants | 24.62 [17.49 to 32.94] | 9.23 [3.46 to 19.02]
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Superiority; p = 0.0095, Cochran-Mantel-Haenszel; Stratified Cochran-Mantel-Haenszel = 15.67, 95% CI 2-sided [5.54 to 25.81]

2. Secondary Outcome: Percentage of Participants With Transfusion Independence (TI) at Week 24
Description: TI status was defined as not receiving red blood cell (RBC) or whole blood transfusion for >=12 weeks, with no hemoglobin (Hgb) level < 8 grams per deciliter (g/dL) during the same interval. Percentage of participants with TI have been presented.
Time Frame: Week 24
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Percentage of Participants | 30.0 [22.28 to 38.66] | 20.00 [11.10 to 31.77]
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Non-Inferiority — If the lower bound of the confidence interval (CI) is greater than 0, MMB was to be declared non-inferior to DAN; p = 0.0116, Cochran-Mantel-Haenszel; Non-inferiority difference = 13.58, 95% CI 2-sided [1.86 to 25.30] — Non-inferiority difference, defined as p(MMB) - (0.8) *p(DAN) where p(MMB) is percentage of participants with TI status in MMB arm and p(DAN) is percentage of participants with TI status in DAN arm

3. Secondary Outcome: Splenic Response Rate (SRR) of >=25% at Week 24
Description: Splenic response rate (SRR) is defined as the percentage of participants who have reduction in spleen volume of >=25% from Baseline at the end of Week 24. Baseline was the last assessment done before or on the day of first dose date.
Time Frame: Baseline and Week 24
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Percentage of Participants | 39.23 [30.79 to 48.18] | 6.15 [1.70 to 15.01]
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified Cochran-Mantel-Haenszel = 33.05, 95% CI 2-sided [22.59 to 43.51]

4. Secondary Outcome: Change From Baseline in MFSAF TSS at Week 24
Description: TSS was measured using the MFSAF v4.0. The MFSAF v4.0 comprises 7 domains representing the 7 most relevant symptoms of MF identified through existing participant and clinician-based evidence: fatigue, night sweats, pruritus, abdominal discomfort, pain under the left ribs, early satiety, and bone pain. Participants scored each symptom domain using an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable). The MFSAF TSS was calculated as the sum of scores of the 7 domains for a possible range of scores of 0 to 70, with a higher TSS corresponding to more severe symptoms. A reduction from Baseline corresponded to a lessening of MF symptoms. Baseline was the last assessment done before or on the day of first dose date. Change from Baseline was defined as the post-Baseline value minus Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Analysis Set. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 92 | 37
Scores on a scale | -9.36 (1.08) | -3.13 (1.62)
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.0014, mixed model for repeated measures (MMRM); Least Squares Mean Difference = -6.22, 95% CI 2-sided [-10.0 to -2.43]

5. Secondary Outcome: Splenic Response Rate (SRR) of >= 35% at Week 24
Description: Splenic response rate (SRR) is defined as the percentage of participants who have reduction in spleen volume of >=35 % from Baseline at the end of Week 24. Baseline was the last assessment done before or on the day of first dose date.
Time Frame: Baseline and Week 24
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Percentage of Participants | 22.31 [15.48 to 30.44] | 3.08 [0.37 to 10.68]
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.0011, Cochran-Mantel-Haenszel; Stratified Cochran-Mantel-Haenszel = 18.18, 95% CI 2-sided [9.77 to 26.59]

6. Secondary Outcome: Percentage of Participants With Zero RBC Units Transfused Over 24-Weeks
Description: Percentage of participants with zero RBC units transfused over 24-weeks were reported.
Time Frame: Up to 24 weeks
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Percentage of participants | 35.38 [27.20 to 44.25] | 16.92 [8.76 to 28.27]
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.0012, Cochran-Mantel-Haenszel; Stratified Cochran-Mantel-Haenszel = 17.20, 95% CI 2-sided [7.99 to 26.40]

7. Secondary Outcome: Percentage of Participants With <=4 RBC Units Transfused Over 24-weeks
Description: Percentage of participants with <=4 RBC units transfused over 24-weeks were reported.
Time Frame: Up to 24 weeks
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Percentage of participants | 55.38 [46.42 to 64.10] | 44.62 [32.27 to 57.47]
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.1133, Cochran-Mantel-Haenszel; Stratified Cochran-Mantel-Haenszel = 10.62, 95% CI 2-sided [-2.40 to 23.64]

8. Secondary Outcome: Duration of MFSAF TSS Response
Description: Duration of MFSAF TSS response is defined as the number of days from the start of the initial 28-day period in which a participant had a >= 50% reduction from Baseline TSS to the first day of the 7-day assessment that determines the mean TSS for the 28-day period during which the participants TSS equals or exceeds their Baseline value.
Time Frame: Up to a maximum of 151 weeks
Population: ITT Analysis Set. Only those participants with data available at specified time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 32 | 6
Days | 286.00 [286.00 to 286.00] | NA [NA to NA] — <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived.

9. Secondary Outcome: Duration of TI Response
Description: Duration of TI is defined as the number of days from (a) the first day of a 12-week period that satisfies the 12-week TI status definition, to (b) the first RBC transfusion or Hgb level < 8 g/dL (except in the case of clinically overt bleeding).
Time Frame: Up to a maximum of 151 weeks
Population: ITT Analysis Set. Only those participants with data available at specified time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 39 | 13
Days | NA [NA to NA] — <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived. | NA [NA to NA] — <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived.

10. Secondary Outcome: Mean Cumulative Number of Whole Blood Units Transfused Over 24 Weeks
Description: Cumulative transfusion risk was calculated as the estimated mean cumulative number of whole blood units transfused during the study.
Time Frame: Up to Week 24
Population: ITT Analysis Set.
Measure: Mean (Standard Deviation); unit: Whole blood units
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Whole blood units | 6.55 (8.413) | 10.86 (13.203)
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.0006, Anderson & Gill proportional means model; Hazard Ratio (HR) = 0.556, 95% CI 2-sided [0.397 to 0.778]

11. Secondary Outcome: Percentage of Participants With Transfusion Dependence (TD) Status at Week 24
Description: TD status at Week 24 is defined as requirement of >=4 RBC units in an 8-week period immediately prior to the end of Week 24.
Time Frame: Week 24
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Percentage of participants | 15.38 [9.66 to 22.76] | 24.62 [14.77 to 36.87]
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.1602, Cochran-Mantel-Haenszel; Stratified CMH = -8.26, 95% CI 2-sided [-20.18 to 3.66]

12. Secondary Outcome: Percentage of Participants With a Hemoglobin Response
Description: Hemoglobin responses are defined as increases of >= 1, >= 1.5, or >= 2 g/dL from Baseline in Hgb, as measured over a (rolling) period of at least 12 consecutive weeks falling entirely before the end of Week 24. Baseline was the last assessment done before or on the day of first dose date. Data has been reported for percentage of participants who had >= 1, >= 1.5, or >= 2 g/dL increase from Baseline in hemoglobin.
Time Frame: Baseline and Week 24
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Percentage of participants
  >=1g/dL Increase | 53.08 [44.13 to 61.88] | 33.85 [22.57 to 46.65]
  >=1.5g/dL Increase | 40.00 [31.51 to 48.95] | 23.08 [13.53 to 35.19]
  >=2g/dL Increase | 29.23 [21.59 to 37.85] | 20.00 [11.10 to 31.77]
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.0124, Cochran-Mantel-Haenszel; Stratified CMH = 19.00, 95% CI 2-sided [4.68 to 33.32] — >=1g/dL Increase in Hemoglobin response
Statistical Analysis 2: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.0282, Cochran-Mantel-Haenszel; Stratified CMH = 15.68, 95% CI 2-sided [2.47 to 28.90] — >=1.5g/dL Increase in Hemoglobin response
Statistical Analysis 3: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.2844, Cochran-Mantel-Haenszel; Stratified CMH = 6.97, 95% CI 2-sided [-5.41 to 19.35] — >=2g/dL Increase in Hemoglobin response

13. Secondary Outcome: Number of Baseline TD Participants With TI Status at Week 24
Description: Participants were defined as having TD if they met both of the following requirements in the 8 weeks immediately before the end of Week 24: >= 4 red blood cell or whole blood units were transfused (except in the case of clinically overt bleeding), each in response to a hemoglobin assessment of <= 9.5 g/dL; and there were >= 2 hemoglobin assessments with >= 28 days between the earliest and latest hemoglobin assessments. TI status was defined as not requiring red blood cell transfusion (except in the case of clinically overt bleeding) for >= 12 weeks immediately prior to the end of Week 24, with hemoglobin levels >= 8 g/dL.
Time Frame: Week 24
Population: ITT Analysis Set. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 63 | 34
Participants | 9 | 3

14. Secondary Outcome: Duration of TI in Baseline TD Participants
Description: as for outcome 9
Time Frame: Up to a maximum of 151 weeks
Population: ITT Analysis Set. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 63 | 34
Days | NA [224.0 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived | NA [196.0 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived.

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs)- up to Week 24
Description: An adverse event (AE) is any untoward medical occurrence in a trial participant administered an investigational product(s), a comparator product, or an approved drug regardless of the causal relationship with treatment. An SAE is an AE that Results in death, life threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, results in a congenital anomaly/birth defect or any important medical events as per medical or scientific judgment. Adverse events which were not Serious were considered as Non-Serious adverse events.
Time Frame: Up to Week 24
Population: Safety analysis set included all participants in the ITT Analysis set who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- MMB 200 mg QD + Placebo- Randomized Double-Blind Treatment Period: Participants were randomized to receive 200 mg of MMB orally QD and a DAN-placebo orally BID during the randomized 24-week double-blind treatment period.
- DAN 300 mg BID + Placebo- Randomized Double-Blind Treatment Period: Participants were randomized to receive 300 mg of DAN orally BID and MMB-placebo orally QD during the randomized 24-week double-blind treatment period.
Arm/Group | MMB 200 mg QD + Placebo- Randomized Double-Blind Treatment Period | DAN 300 mg BID + Placebo- Randomized Double-Blind Treatment Period
Number analyzed (Participants) | 130 | 65
Participants
  Any non-SAEs | 108 | 55
  Any SAEs | 45 | 26

16. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs)- From Week 24 to a Maximum of 151 Weeks
Description: An AE is any untoward medical occurrence in a trial participant administered an investigational product(s), a comparator product, or an approved drug regardless of the causal relationship with treatment. An SAE is an AE that Results in death, life threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, results in a congenital anomaly/birth defect or any important medical events as per medical or scientific judgment. Adverse events which were not Serious were considered as Non-Serious adverse events.
Time Frame: From Week 24 to a maximum of 151 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- MMB 200 mg QD- Open-Label Extended Treatment Period: Participants who completed the randomized treatment period or discontinued treatment early for other reasons but completed scheduled assessments through Week 24 were enrolled in an open-label extended treatment period. Participants continued to receive 200 mg of MMB orally QD during the open-label extended treatment period.
- DAN 300 mg BID to MMB 200 mg QD- Open-Label Extended Treatment Period: Participants who completed the randomized treatment period, discontinued treatment early due to splenic progression, or discontinued treatment early for other reasons but completed scheduled assessments through Week 24 were enrolled in an open-label extended treatment period. Participants who received DAN 300 mg BID during randomized period switched to receive 200 mg of MMB orally QD during open-label extended treatment period.
Arm/Group | MMB 200 mg QD- Open-Label Extended Treatment Period | DAN 300 mg BID to MMB 200 mg QD- Open-Label Extended Treatment Period
Number analyzed (Participants) | 93 | 41
Participants
  Any non-SAEs | 57 | 28
  Any SAEs | 30 | 12

17. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the interval from the first study drug dosing date (or randomization date for participants who did not receive treatment) to death from any cause.
Time Frame: Up to a maximum of 151 weeks
Population: ITT Analysis Set. Values are presented based on the Kaplan-Meier analysis. All participants (overall population) were included in analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Days | 624.0 [333.0 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | NA [309.00 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.6879, Log Rank; Hazard Ratio (HR) = 0.890, 95% CI 2-sided [0.504 to 1.572]

18. Secondary Outcome: Leukemia-free Survival (LFS)
Description: LFS is defined as the interval from first study drug dosing date (or randomization date for participants who did not receive treatment) to any evidence of leukemic transformation and/or death (from any cause).
Time Frame: Up to a maximum of 151 weeks
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 130 | 65
Days | 624.0 [325.0 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived | NA [284.0 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived.
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.4320, Log Rank; Hazard Ratio (HR) = 0.804, 95% CI 2-sided [0.466 to 1.386]

19. Secondary Outcome: Change From Baseline in Disease-related Fatigue as Assessed by MFSAF TSS v4.0 at Week 24
Description: The MFSAF v4.0 comprises 7 domains representing the 7 most relevant symptoms of MF identified through existing participant- and clinician-based evidence: fatigue, night sweats, pruritus, abdominal discomfort, pain under the left ribs, early satiety, and bone pain. Participants scored each symptom domain using an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable). Data has been reported for Disease-related Fatigue domain measured using an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable), higher score indicates worst outcome. An increase in score from Baseline indicated a worsening of fatigue and a decrease in score from Baseline indicated an improvement in fatigue. Baseline was the last assessment done before or on the day of first dose date. Change from Baseline was defined as the post-Baseline value minus Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Analysis Set. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 92 | 37
Scores on a scale | -1.53 (0.20) | -0.82 (0.31)
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.0513, MMRM; Least Squares Mean Difference = -0.71, 95% CI 2-sided [-1.42 to 0.00]

20. Secondary Outcome: Change From Baseline in Cancer-related Fatigue as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) at Week 24
Description: The EORTC QLQ-C30 is comprised of 5 functional scales (physical, role, emotional, social, cognitive), eight single item symptom scales (fatigue, pain, nausea/vomiting, appetite loss, constipation, diarrhea, insomnia, dyspnea), as well as sub-scales assessing global health/quality of life and financial impact. Most items use a 4-point Likert scale from "not at all" to "very much" and a one-week recall period with the exception of the final two items which use a 7 point scale response from "very poor" to "excellent". Scores were averaged and transformed to a 0-100 scale, with higher scores representing better functioning/quality of life. An increase in scores from Baseline indicated an improved functioning/quality of life, and a decrease in scores from Baseline indicated a worsened functioning/quality of life. Baseline was the last assessment done before or on the day of first dose date. Change from Baseline was defined as the post-Baseline value minus Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Analysis Set. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 89 | 35
Scores on a scale | -14.34 (2.35) | -3.52 (3.65)
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.0113, MMRM; Least Squares Mean Difference = -10.82, 95% CI 2-sided [-19.15 to -2.48]

21. Secondary Outcome: Change From Baseline in Physical Function Score as Assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 10b at Week 24
Description: PROMIS Physical Function Short Form 10b consists of 14 questions; each with a 5-point response. PROMIS short form assesses self-reported capability of a participant rather than actual performance of physical activities. This includes functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back) as well as instrumental activities of daily living, such as running errands. Participants scored each response on a scale from 1 (unable to do) to 5 (without any difficulty, or not at all). Total possible range of scores was 14 to 70, with higher scores corresponding to a greater physical function ability. An increase in score from Baseline indicated an improvement in physical function ability and a decrease in score from Baseline indicated a reduction in physical function ability. Baseline was last assessment done before or on the day of first dose date. Change from Baseline was defined as post-Baseline value minus Baseline value.
Time Frame: Baseline and Week 24
Population: ITT Analysis Set. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | MMB 200 mg QD + Placebo | DAN 300 mg BID + Placebo
Number analyzed (Participants) | 89 | 32
Scores on a scale | 1.19 (0.77) | -0.11 (1.21)
Statistical Analysis 1: Comparison: MMB 200 mg QD + Placebo vs DAN 300 mg BID + Placebo; Test type: Other; p = 0.3570, MMRM; Least Squares Mean Difference = 1.31, 95% CI 2-sided [-1.49 to 4.11]

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs) and non-SAEs were collected up to Week 24 for Randomized Double-Blind Treatment Period and From Week 24 to a maximum of 151 weeks for the Open-Label Extended Treatment Period
Description: Serious adverse events (SAEs) and non-SAEs were measured in the Safety analysis set, which included all participants in the ITT analysis set who received at least one dose of study drug. All-cause mortality was measured in the ITT analysis set, which included all randomized participants. Data are presented per treatment received.
Arm/Group | MMB 200 mg QD + Placebo- Randomized Double-Blind Treatment Period | DAN 300 mg BID + Placebo- Randomized Double-Blind Treatment Period | MMB 200 mg QD- Open-Label Extended Treatment Period | DAN 300 mg BID to MMB 200 mg QD- Open-Label Extended Treatment Period
All-Cause Mortality (participants affected / at risk) | 25/130 | 16/65 | 23/93 | 8/41
Serious Adverse Events (participants affected / at risk) | 45/130 | 26/65 | 30/93 | 12/41
Other Adverse Events (participants affected / at risk) | 108/130 | 55/65 | 57/93 | 28/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMB 200 mg QD + Placebo- Randomized Double-Blind Treatment Period (N=130) | DAN 300 mg BID + Placebo- Randomized Double-Blind Treatment Period (N=65) | MMB 200 mg QD- Open-Label Extended Treatment Period (N=93) | DAN 300 mg BID to MMB 200 mg QD- Open-Label Extended Treatment Period (N=41)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 1 (1) | 1 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Listeria sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 6 (6) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (6) | 3 (3) | 2 (2) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMB 200 mg QD + Placebo- Randomized Double-Blind Treatment Period (N=130) | DAN 300 mg BID + Placebo- Randomized Double-Blind Treatment Period (N=65) | MMB 200 mg QD- Open-Label Extended Treatment Period (N=93) | DAN 300 mg BID to MMB 200 mg QD- Open-Label Extended Treatment Period (N=41)
Anaemia (Blood and lymphatic system disorders) | 12 (34) | 6 (11) | 9 (18) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 7 (11) | 2 (5) | 5 (9) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 28 (50) | 7 (11) | 13 (22) | 7 (10)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 6 (6) | 3 (3) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 5 (6) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (13) | 5 (5) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 29 (40) | 6 (7) | 16 (21) | 5 (7)
Nausea (Gastrointestinal disorders) | 21 (28) | 6 (6) | 8 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (10) | 0 (0) | 3 (3) | 1 (1)
Asthenia (General disorders) | 17 (20) | 6 (8) | 12 (15) | 0 (0)
Fatigue (General disorders) | 8 (10) | 6 (10) | 6 (11) | 3 (3)
Oedema peripheral (General disorders) | 9 (9) | 9 (10) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 11 (13) | 5 (6) | 12 (13) | 3 (4)
COVID-19 (Infections and infestations) | 9 (9) | 0 (0) | 8 (8) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (9) | 3 (3) | 4 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (13) | 5 (11) | 2 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (9) | 4 (5) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 10 (18) | 0 (0) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 10 (18) | 10 (16) | 7 (13) | 4 (4)
Platelet count decreased (Investigations) | 9 (24) | 3 (4) | 3 (7) | 1 (2)
Weight decreased (Investigations) | 14 (16) | 3 (4) | 9 (9) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 9 (13) | 6 (8) | 4 (5) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (7) | 6 (12) | 2 (3) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (9) | 4 (6) | 3 (3) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (5) | 4 (4) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 8 (9) | 1 (1) | 1 (1) | 4 (4)
Paraesthesia (Nervous system disorders) | 8 (10) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (2) | 8 (9) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 10 (12) | 7 (8) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (6) | 1 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (14) | 7 (7) | 6 (7) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 6 (6) | 3 (3) | 5 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GlaxoSmithKline (GSK) agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04173494/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT04173494/SAP_001.pdf